CLINICAL TRIAL: NCT01831687
Title: An Open Label, Balanced, Randomized, Single-dose, Two-treatment, Two-sequence, Two-period, Crossover, Oral Bioequivalence Study of Etodolac Extended Release Tablets USP 600mg of Ipca Laboratories Limited, India and Etodolac Extended Release Tablets 600mg of Teva Pharmaceutical Ind. Ltd., USA in Healthy, Adult, Human Subjects Under Fed Condition
Brief Title: Bioequivalence Study of Etodolac Extended Release Tablets USP 600mg Under Fed Condition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: IPCA Laboratories Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Ipca/11-VIN-414
Record Dates: First submitted 2013-04-06; First posted 2013-04-15 (Estimated); Last update posted 2013-04-15 (Estimated); Status verified 2013-04

CONDITIONS: Fasting
MeSH Terms: conditions — Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Etodolac Extended Release Tablets 600mg (Active Comparator): Etodolac Extended Release Tablets 600mg of Teva Pharmaceutical Ind. Ltd., USA
  Interventions: Drug: Etodolac Extended Release Tablets USP 600mg; Drug: Etodolac Extended Release Tablets 600mg
- Etodolac Extended Release Tablets USP 600mg (Experimental): Etodolac Extended Release Tablets USP 600mg of Ipca Laboratories Limited, India
  Interventions: Drug: Etodolac Extended Release Tablets USP 600mg; Drug: Etodolac Extended Release Tablets 600mg

INTERVENTIONS:
Drug: Etodolac Extended Release Tablets USP 600mg — Etodolac Extended Release Tablets USP 600mg once a day
  Other Names: Test product
Drug: Etodolac Extended Release Tablets 600mg — Etodolac Extended Release Tablets 600mg once a day
  Other Names: Reference product

SUMMARY:
This is a open Label, balanced, randomized, single dose, two-treatment, two-sequence, two-period, crossover, oral pivotal bioequivalence study. The purpose of this study is to assess the bioequivalence between Test Product and the corresponding Reference Product under fed condition in healthy, adult human subjects.

DETAILED DESCRIPTION:
Objective of this pivotal study was to assess the bioequivalence between Test Product: Etodolac Extended Release Tablets USP 600mg of Ipca Laboratories Limited, India and the corresponding Reference Product: Etodolac Extended Release Tablets 600 mg of Teva Pharmaceutical Ind. Ltd., USA under fed condition in healthy, adult, human subjects in a randomized crossover study.

The study was conducted with 36 healthy adult subjects. In each study period, a single 600 mg dose of either test or reference was administered to the subjects as per the randomization schedule in each study period with about 240 mL of water at ambient temperature in sitting position.

The duration of the clinical phase was approximately 15 days including washout period of 11 days between administrations of study drug in each study period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and non-pregnant female subjects (age range of 18 to 45 years).
* Body Mass Index (18.5 to 24.9 kg/m2) with minimum of 50 kg weight.
* Subjects with normal health as determined by personal medical and medication history, clinical examination and laboratory examinations within the clinically acceptable reference range.
* Subjects having normal 12-lead electrocardiogram (ECG)and normal chest X-Ray (P/A view).
* Subjects having negative urine screen for drugs of abuse (including amphetamines, barbiturates, benzodiazepines, marijuana, cocaine, and morphine).
* Subjects having negative alcohol breath test.
* Subjects willing to adhere to protocol requirements and to provide written informed consent.
* Subjects having negative beta-hCG Pregnancy test (only for female subjects).
* For Female Subjects:
* Female of child bearing potential practicing an acceptable method of birth control for the duration of the study as judged by the investigator(s), such as condoms, foams, jellies, diaphragm, intrauterine device (IUD), or abstinence, or
* Postmenopausal for at least 1 years, or if less than 1 years, then following acceptable contraceptive measures as mentioned above
* Surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy has been performed on the subject).

Exclusion Criteria:

* Hypersensitivity to Etodolac or related class of drugs.
* History or presence of significant cardiovascular, pulmonary, hepatic, renal, gastrointestinal, endocrine, immunological, dermatological, neurological or psychiatric disease or disorder.
* History or presence of significant alcoholism or drug abuse.
* History or presence of significant smoking.
* History or presence of significant asthma, urticaria or other allergic reactions.
* History or presence of significant gastric and/or duodenal ulceration.
* History or presence of significant thyroid disease, adrenal dysfunction, organic intracranial lesion such as pituitary tumor.
* History or presence of cancer.
* Difficulty with donating blood.
* Difficulty in swallowing solids like tablets or capsules.
* Use of any prescribed medication or OTC medical products during last two weeks prior to dosing in period 01.
* Major illness during 3 months before screening.
* Participation in a drug research study within past 3 months.
* Donation of blood in the past 3 months before screening.
* Consumption of grapefruit juice, xanthine-containing products, tobacco containing products or alcohol within 48 hours prior to dosing.
* Positive screening test for any one or more: HIV, Hepatitis B and Hepatitis C.
* History or presence of significant easy bruising or bleeding.
* History or presence of significant recent trauma.
* Subjects who have been on an abnormal diet (for whatever reason) during the four weeks preceding the study.
* Female subjects who are currently on breast feeding.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2012-12; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Bioequivalence is based on Cmax and AUC parameters. | 1 Months
  Sampling hours: Pre-dose and at 1.00, 2.00, 3.00, 3.50, 4.00, 4.50, 5.00, 5.50, 6.00, 6.50, 7.00, 7.50, 8.00, 9.00, 10.00, 12.00, 16.00, 24.00, 36.00 and 48.00 hours post dose.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Hardik Dave, M.B.B.S, Principal Investigator — Veeda Clinical Research Pvt. Ltd.
Locations (1):
- Veeda Clinical Research Pvt. Ltd., Ahmedabad, Gujarat, India